CLINICAL TRIAL: NCT03960008
Title: A Randomized Multi-Center Phase III Study of Individualized Stereotactic Body Radiation Therapy (SBRT) Versus Trans-Arterial Chemoembolization (TACE) as a Bridge to Transplant in Hepatocellular Carcinoma.
Brief Title: Stereotactic Body Radiation Therapy (SBRT) vs Trans-Arterial Chemoembolization (TACE) as Bridge to Transplant
Acronym: SBRTvsTACE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was closed early due to lack of enrollments and insufficient funding.
Sponsor: Lahey Clinic (Other)
Collaborators: Varian Medical Systems (Industry); Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20193013
Record Dates: First submitted 2019-04-30; First posted 2019-05-22 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma; HCC
Keywords: Hepatocellular Carcinoma (HCC); Liver transplant; Bridge to transplant; Stereotactic body radiation therapy (SBRT); Trans-arterial chemoembolization (TACE)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; Radiotherapy; Chemoembolization, Therapeutic; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Stereotactic Body Radiation Therapy (SBRT) (Other): Radiation Therapy
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Trans-Arterial Chemoembolization (TACE) (Other): Procedure/Surgery - Chemoembolization Drug: Doxorubin
  Interventions: Procedure: Trans-Arterial Chemoembolization (TACE); Drug: Doxorubin

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT will be delivered in five total fractions, with at a minimum of one day between any two treatments. The entire treatment must be delivered within 15 total days.
  Other Names: Radiation Therapy
  Arms: Stereotactic Body Radiation Therapy (SBRT)
Procedure: Trans-Arterial Chemoembolization (TACE) — First day will be administered and a second TACE will be administered after 4 weeks and subsequently if imaging is showing disease progression. Following each TACE procedure all patients will remain in hospital for observation
  Other Names: Chemoembolization
  Arms: Trans-Arterial Chemoembolization (TACE)
Drug: Doxorubin — This procedure will be completed with 2 vials of drug eluting beads each loaded with 50 mg of Doxorubin.
  Other Names: Doxorubin bead therapy
  Arms: Trans-Arterial Chemoembolization (TACE)

SUMMARY:
This study will compare stereotactic body radiation therapy (SBRT) to trans-arterial chemoembolization (TACE) as a bridging strategy for patients with HCC undergoing liver transplantation. We propose that SBRT will be associated with longer time intervals between initial treatment and the need for retreatment, compared to TACE, as a "bridge" to liver transplantation in subjects with HCC.

DETAILED DESCRIPTION:
For patients with hepatocellular carcinoma (HCC) who are waiting for a liver transplant, local treatment of their disease has become the standard of care in an effort to decrease dropout rates and as a means of reducing tumor recurrence after transplantation. For patients undergoing local regional therapy as a bridge to transplantation, trans-arterial chemoembolization (TACE) is the most commonly utilized treatment. However, the best modality for patients undergoing treatment as a bridge to transplantation is unclear. A newer strategy for the treatment of HCC is stereotactic body radiation therapy (SBRT). This study will compare SBRT to TACE as a bridging strategy for patients with HCC undergoing liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with HCC are eligible for this trial. HCC is defined as having at least one of the following:

   * Biopsy proven HCC or:
   * A discrete hepatic tumor(s) as defined by the Barcelona (29) criteria for cirrhotic subjects, ≥2cm with arterial hypervascularity and venous or delayed phase washout on CT or MRI.
2. Subjects are liver transplant candidates (actively awaiting organ transplant per transplant services in documentation), or, potential liver transplant candidates (at the discretion of the liver team and/or Principal Investigator) advised by liver transplant services as needing local treatment prior to liver transplant evaluation.
3. Subjects must be within UCSF criteria (one solitary tumor smaller than 6.5 cm, or patients having 3 or fewer nodules, with the largest lesion being smaller than 4.5 cm or having a total tumor diameter less than 8.5 cm without vascular invasion) and eligible for potential liver transplant.
4. Subjects must be eligible per standard of care for either TACE or SBRT procedures.
5. Subjects must have a life expectancy of at least 12 weeks.
6. Subjects must be 18 years of age or older. Adult subjects of all ages, both sexes and all races will be included in this study.
7. Subjects must sign an informed consent form approved for this purpose by the Institutional Review Board (IRB) of record .
8. Subjects must have a Child-Turcotte-Pugh (CTP) score ≤8.
9. Patients must have adequate organ function within 2 weeks of enrollment.

   * Bone marrow: Platelets ≥30,000/mm3
   * Renal: BUN ≤40 mg/dl; creatinine ≤2.0 mg/dl
   * Hepatic: INR ≤ 1.5 or correctable by Vitamin K, unless anti-coagulated for another medical reason
   * Bilirubin < 3.0 mg/dl (in the absence of obstruction or pre-existing disease of the biliary tract, e.g. primary sclerosing cholangitis).
10. Patients uninvolved liver volume will be estimated and must be > 700ml.
11. Patients must have a Zubrod performance status of ≤2.

Exclusion Criteria:

1. Subjects in a "special category" designated by the Public Health Service, Including subjects younger than 18, pregnant women, and prisoners.
2. Refractory ascites that requires paracentesis for management.
3. Known allergy to intravenous iodinated contrast agents unresponsive to prednisone pre-treatment.
4. History of prior radiation to the liver.
5. Evidence of metastatic disease.
6. Presence of a Trans-jugular intra-hepatic porto-systemic shunt (TIPS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corrine Zarwan, MD, Principal Investigator — Lahey Hospital & Medical Center
Locations (5):
- United States (4):
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
- Princess Margaret Hospital, UHN, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) | Trans-Arterial Chemoembolization (TACE)
Started | 4 | 5
Completed | 0 | 0
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) | Trans-Arterial Chemoembolization (TACE) | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (3.9) | 60.6 (7.6) | 62.8 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 1 | 2
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: To Compare the Duration of Disease Control in Treated Lesions When Utilizing SBRT Versus TACE as a Bridging Strategy for Patients With HCC Eligible for Liver Transplantation
Description: To compare whether or not there was disease present in treated lesions in both the SBRT and TACE arms in patients eligible for liver transplant at 1 year post treatment.
Time Frame: 1 year post treatment
Population: Data has not been collected and therefore not analyzed for this outcome.
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) | Trans-Arterial Chemoembolization (TACE)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Compare Participants With Treatment-related Adverse Events as Assessed by CTCAE v5.0
Description: To compare treatment related adverse events between both arms, SBRT and TACE.
Time Frame: At each treatment, 2 weeks post treatment, 2 months post treatment, 5 months post treatment, every 3 months until 24 months post treatment
Population: Data has not been collected and therefore not analyzed for this outcome
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) | Trans-Arterial Chemoembolization (TACE)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Further Interventions
Description: To compare the number of further interventions between the SBRT and TACE arms.
Time Frame: 2 weeks post treatment, 2 months post treatment, 5 months post treatment, every 3 months until 24 months post treatment
Population: Data has not been collected and therefore not analyzed for this outcome.
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) | Trans-Arterial Chemoembolization (TACE)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Rate of Pathological Response of Treated Lesion(s)
Description: Complete pathologic response of lesions will be analyzed on the explant liver specimen after liver transplant. The pathology note will be consulted.
Time Frame: Review of pathology report after liver transplant
Population: Data has not been collected and therefore not analyzed for this outcome.
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) | Trans-Arterial Chemoembolization (TACE)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Rate of Radiological Response of Treated Lesion(s)
Description: Response of treated lesions will be analyzed at protocol specified time frames. The response rate between both treatment arms will be compared.
Time Frame: Baseline, 2 months post-treatment, 5 months post-treatment, every 3 months thereafter until 2 years post treatment
Population: Data has not been collected and therefore not analyzed for this outcome
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) | Trans-Arterial Chemoembolization (TACE)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: To Assess Quality of Life by Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) Questionnaire
Description: A 45-item self-report instrument to measure health-related quality of life (HRQL) in patients with hepatobiliary cancers and is one of the most widely-used instruments in this clinical area. The FACT-Hep consists of the 27-item FACT-G, assesses HRQL, and the 18-item Hepatobiliary Subscale (HS), assesses disease-specific issues such as pain, appetite, and cramping. The FACT-G evaluates physical well-being, social/family well-being, emotional well-being, and functional well-being. Sections have a 7-day reference period and are scored from 0-4 ("not at all" to "very much"), with higher scores indicating better HRQL. Score ranges are 0-28 for physical well-being, 0-28 for social/family well-being, 0-24 for emotional well-being, 0-28 for functional well-being, and 0-72 for the HS. All subscale scores from the FACT-G and HS can be summed together to create a total FACT-Hep score, with a possible range of 0-180. The FACT-Hep takes approximately 10 minutes to complete.
Time Frame: Baseline, during treatment, 2 months post-treatment, 5 months post-treatment, every 3 months until 24 months post treatment
Population: Data has not been collected and therefore not analyzed for this outcome.
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) | Trans-Arterial Chemoembolization (TACE)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: To Assess Over Survival
Description: Overall survival will be compared in both arms at protocol specified time frames.
Time Frame: as for outcome 6
Population: Data has not been collected and therefore not analyzed for this outcome
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) | Trans-Arterial Chemoembolization (TACE)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: To Assess 90 Day Post-transplant Morbidity
Description: Compare the morbidity at 90 days post transplant between both arms.
Time Frame: Disease status to be captured 90 days post-transplantation (+/- 2 weeks)
Population: Data has not been collected and therefore not analyzed for this outcome
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) | Trans-Arterial Chemoembolization (TACE)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: To Assess 90 Day Post-transplant Mortality
Description: Will assess the mortality of post-transplant patients between the two arms.
Time Frame: Survival status to be captured 90 days post-transplantation (+/- 2 weeks)
Population: Data has not been collected and therefore not analyzed for this outcome.
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) | Trans-Arterial Chemoembolization (TACE)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline, During Treatment, post treatment follow-up visit, 3 Month, 6 Month, then every 3 months until 24 month time point.
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) | Trans-Arterial Chemoembolization (TACE)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
This study closed to accrual early, with the limited number of participants, we were unable to analyze the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT03960008/Prot_SAP_001.pdf